CLINICAL TRIAL: NCT00360399
Title: Predictors of Antidepressant Treatment Response: The Emory CIDAR
Brief Title: Identifying Factors That Predict Antidepressant Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Mayberg, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00024975; P50MH077083 (NIH)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Depression
Keywords: Escitalopram; Duloxetine; Cognitive Behavioral Therapy; PET; fMRI
MeSH Terms: conditions — Depression | interventions — Escitalopram; Duloxetine Hydrochloride; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Escitalopram (Active Comparator): Participants will receive treatment with escitalopram for 12 weeks
  Interventions: Drug: Escitalopram
- Duloxetine (Active Comparator): Participants will receive treatment with duloxetine for 12 weeks
  Interventions: Drug: Duloxetine
- CBT (Active Comparator): Participants will receive 16 one-hour sessions of cognitive behavioral therapy delivered over 12 weeks
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 to 20 mg per day for 12 weeks
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Duloxetine — Duloxetine 30 to 60 mg per day for 12 weeks
  Other Names: Cymbalta
  Arms: Duloxetine
Behavioral: Cognitive behavioral therapy (CBT) — CBT will include 16 one-hour sessions provided over 12 weeks.
  Arms: CBT

SUMMARY:
This study will compare different treatments for depression in order to identify which factors predict effectiveness, and will include a companion study which investigates combining treatments and long term effectiveness.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a serious illness that affects a person's body, mood, and thoughts. The symptoms of MDD can interfere with a person's ability to work, study, sleep, eat, and enjoy activities that were once pleasurable. Antidepressant medications and psychotherapy are among the effective treatments for MDD. Individuals often respond to one type of treatment, but not another. Currently, however, doctors have no way of pre-determining which individuals will most benefit from which treatments. In the absence of practical predictors of MDD treatment response, the potential efficacy of existing MDD treatments is limited. This study will identify factors that may predict MDD treatment response by comparing the effectiveness of a selective serotonin reuptake inhibitor (SSRI), a serotonin norepinephrine reuptake inhibitor (SNRI), and cognitive behavioral therapy in people with MDD.

Participants in this 14-week, double-blind study will be randomly assigned to receive duloxetine (SNRI), escitalopram (SSRI), or cognitive behavioral therapy. During the first 2 weeks of screening, participants will complete questionnaires, clinician evaluations, an electrocardiogram, a personality assessment, a dexamethasone-corticotropin releasing factor test, a functional magnetic resonance imaging scan and provide blood samples. Upon completion of screening, patients will start the treatment to which they were randomized. Duloxetine and escitalopram are two medications that are approved by the Food and Drug Administration for the treatment of depression. Cognitive behavioral therapy is a talking therapy that is also used to treat depression. All participants assigned to take duloxetine or escitalopram will be seen by a study physician weekly for 6 weeks, and then every other week for the remainder of the study. Participants assigned to cognitive behavioral therapy will attend therapy sessions twice a week for the first 4 weeks, and then once a week for the remainder of the study. The following assessments will be performed for all participants at each visit: vital sign and weight measurements; clinician assessments; and self-report questionnaires. Additionally, blood samples will be taken at three visits through the trial and functional magnetic resonance imaging (fMRI) scans will be performed at selected times.

A companion study to the main CIDAR study offers participants further treatment. Participants who achieve remission after the initial 12 weeks of treatment will have the option to enroll in a 21-month follow-up study of maintenance treatment, with visits every three months to monitor for sustained response and relapse. Participants who do not remit will have the option to enroll in another 12-week treatment course, receiving a combination of CBT and medication. Participants who achieve response after this combination treatment will be eligible to receive maintenance combination treatment for up to an additional 18 months, monitored for sustained response and relapse. Participants who do not wish to enroll or continue in the companion study will be provided with a referral for treatment with another mental health provider.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV diagnosis of major depressive episode, as determined by Structured Clinical Interview for DSM-IV (SCID-IV)
* Primary diagnosis of MDD, based on prominence of symptoms and target for intervention (comorbid anxiety disorders, except obsessive-compulsive disorder (OCD), will not be criteria for exclusion)
* Score of at least 18 on the 17-item Hamilton Rating Scale for Depression (HAM-D17)
* Agrees to use an effective form of contraception and/or double barrier method

Exclusion Criteria:

* Previously treated for major depression with either medication or psychotherapy
* Current psychosis, dementia, eating disorder, or dissociative disorder
* History of bipolar disorder (I and II) or schizophrenia
* Alcohol or drug dependence within 3 months prior to study entry or current alcohol or drug abuse (excluding nicotine and caffeine), as assessed by medical history and urine drug screening
* Requires neuroleptic or mood stabilizer therapy in addition to depression treatment
* Presence of any acute or chronic medical disorder that could affect successful completion of the trial
* Medical contraindications that would preclude treatment with escitalopram or duloxetine
* Presence of practical issues that would likely prevent completion of the study (e.g., planned geographical relocation)
* Pregnant or breastfeeding
* Medical conditions that could prevent the safe use of MRI (e.g., pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, or other implants; steel worker)
* Medical conditions that could prevent the safe completion of a dexamethasone-corticotropin releasing factor (Dex-CRF) test (e.g., uncontrolled hypertension, significant abnormalities in EKG, anemia, known allergies against drugs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2006-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen S. Mayberg, MD, Principal Investigator — Emory University; W. Edward Craighead, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Mood and Anxiety Disorders Program, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia

REFERENCES:
- [Background] Dunlop BW, Binder EB, Cubells JF, Goodman MM, Kelley ME, Kinkead B, Kutner M, Nemeroff CB, Newport DJ, Owens MJ, Pace TW, Ritchie JC, Rivera VA, Westen D, Craighead WE, Mayberg HS. Predictors of remission in depression to individual and combined treatments (PReDICT): study protocol for a randomized controlled trial. Trials. 2012 Jul 9;13:106. doi: 10.1186/1745-6215-13-106. PMID 22776534
- [Derived] Dunlop BW, Cha J, Choi KS, Rajendra JK, Nemeroff CB, Craighead WE, Mayberg HS. Shared and Unique Changes in Brain Connectivity Among Depressed Patients After Remission With Pharmacotherapy Versus Psychotherapy. Am J Psychiatry. 2023 Mar 1;180(3):218-229. doi: 10.1176/appi.ajp.21070727. Epub 2023 Jan 18. PMID 36651624
- [Derived] Brydges CR, Fiehn O, Mayberg HS, Schreiber H, Dehkordi SM, Bhattacharyya S, Cha J, Choi KS, Craighead WE, Krishnan RR, Rush AJ, Dunlop BW, Kaddurah-Daouk R; Mood Disorders Precision Medicine Consortium. Indoxyl sulfate, a gut microbiome-derived uremic toxin, is associated with psychic anxiety and its functional magnetic resonance imaging-based neurologic signature. Sci Rep. 2021 Oct 25;11(1):21011. doi: 10.1038/s41598-021-99845-1. PMID 34697401
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Kennedy JC, Dunlop BW, Craighead LW, Nemeroff CB, Mayberg HS, Craighead WE. Follow-up of monotherapy remitters in the PReDICT study: Maintenance treatment outcomes and clinical predictors of recurrence. J Consult Clin Psychol. 2018 Feb;86(2):189-199. doi: 10.1037/ccp0000279. PMID 29369664
- [Derived] Dunlop BW, Rajendra JK, Craighead WE, Kelley ME, McGrath CL, Choi KS, Kinkead B, Nemeroff CB, Mayberg HS. Functional Connectivity of the Subcallosal Cingulate Cortex And Differential Outcomes to Treatment With Cognitive-Behavioral Therapy or Antidepressant Medication for Major Depressive Disorder. Am J Psychiatry. 2017 Jun 1;174(6):533-545. doi: 10.1176/appi.ajp.2016.16050518. Epub 2017 Mar 24. PMID 28335622
- See also: Related Info — http://www.emoryclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Emory University Mood and Anxiety Disorders Program. Men and women, aged 18-65, meeting DSM-IV criteria for a current major depressive disorder, and who had not received prior treatment for a mood disorder were eligible. 515 consented to participate in the trial and 344 were randomized to a treatment arm.
Pre-assignment Details: A total of 344 participants were randomized as follows:
  114 randomized to the Escitalopram arm 115 randomized to the Duloxetine arm 115 randomized to the Cognitive behavioral therapy (CBT) arm
  28 participants did not return for a post-randomization assessment, resulting in 316 participants with data to analyze.
Groups:
- Escitalopram: Participants were randomized to receive treatment with escitalopram for 12 weeks, at a dose of 10 to 20 mg per day
- Duloxetine: Participants were randomized to receive treatment with duloxetine for 12 weeks, at a dose of 30 to 60 mg per day
- Cognitive Behavioral Therapy (CBT): Participants were randomized to receive 16 one-hour sessions of cognitive behavioral therapy (CBT) delivered over 12 weeks
Period: Overall Study
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Started | 114 | 115 | 115
Had Post-randomization Assessment | 105 | 106 | 105
Completed | 86 | 79 | 69
Not Completed | 28 | 36 | 46

BASELINE CHARACTERISTICS:
Population: Participants who consented to participate in the trial and who were randomized to a treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT) | Total
Number analyzed (Participants) | 114 | 115 | 115 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 114 | 115 | 115 | 344
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.1) | 38.3 (11.4) | 40.0 (11.3) | 40.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 64 | 196
  Male | 50 | 47 | 51 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 34 | 32 | 102
  Not Hispanic or Latino | 78 | 81 | 83 | 242
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants was categorized as "Caucasian", "Black", and "Other".
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 28 | 23 | 13 | 64
    White | 47 | 56 | 61 | 164
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 39 | 36 | 41 | 116
Region of Enrollment [Number; unit: participants]
  United States | 114 | 115 | 115 | 344
Current Anxiety Disorder [Number; unit: participants]
  Yes | 67 | 67 | 71 | 205
  No | 47 | 48 | 44 | 139
Previous Episode(s) of Depression [Number; unit: participants] — The number of participants who have had 1, 2, or 3 or more prior episodes of depression
  participants
    One | 59 | 51 | 67 | 177
    Two | 20 | 26 | 17 | 63
    Three or more | 33 | 38 | 28 | 99
    None | 2 | 0 | 3 | 5
Chronic Episode of Depression (2 or More Years) [Number; unit: participants] — The number of participants who are experiencing a chronic episode of depression (2 or more years in duration).
  participants
    Yes | 31 | 37 | 38 | 106
    No | 83 | 78 | 77 | 238
History of Suicide Attempt [Number; unit: participants] — The number of participants who have a prior history of suicide attempt.
  participants
    Yes | 4 | 13 | 8 | 25
    No | 110 | 102 | 107 | 319

OUTCOME MEASURES:

1. Primary Outcome: Remission From Major Depressive Episode in Intent to Treat Sample
Description: The percentage of participants who achieved remission from a major depressive episode, using a last observation carried forward (LOCF) dataset, defined as all randomized patients who initiated treatment and had at least one follow-up rating assessment. A score of equal to or greater than 7 on the Hamilton Depression Rating Scale (HDRS) at the last observation was considered to be remission from depression.
Time Frame: Up to 12 Weeks
Population: This population consists of all participants who were randomized and returned for at least one study visit. This population was used for the intent to treat analyses and not all of these individuals completed the study.
Measure: Number; unit: percentage of participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 105 | 106 | 105
percentage of participants | 46.7 | 54.7 | 41.9

2. Primary Outcome: Remission From Major Depressive Episode Among Participants Who Completed the Intervention
Description: The percentage of participants who achieved remission from a major depressive episode. A score of equal to or greater than 7 on the Hamilton Depression Rating Scale (HDRS) after 10 weeks and 12 weeks of the assigned study treatment was considered to be remission from depression.
Time Frame: Measured at Weeks 10 and 12
Population: This population includes participants who completed the trial, per study protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 86 | 79 | 69
percentage of participants | 44.2 | 51.9 | 43.5

3. Secondary Outcome: Number of Participants in Each Category of Response to Treatment of Depressive Symptoms, in Intent to Treat Sample
Description: Four mutually exclusive categorical outcomes were defined based on the last valid Hamilton Depression Rating Scale (HDRS) rating at the last observation:
  1. Non-response: <30% reduction from baseline
  2. Partial Response: 30-49% reduction from baseline
  3. Response without remission: ≥50% reduction from baseline, but HDRS-17 score >7
  4. Remission: HDRS score ≤7
Time Frame: Up to 12 Weeks
Population: The population is defined as all randomized patients who initiated treatment and had at least one follow-up rating assessment.
Measure: Number; unit: participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 105 | 106 | 105
participants
  Non-Response | 26 | 21 | 32
  Partial Response | 12 | 16 | 19
  Response without remission | 18 | 11 | 10
  Remission | 49 | 58 | 44

4. Secondary Outcome: Number of Participants in Each Category of Response to Treatment of Depressive Symptoms, Among Participants Who Completed the Intervention
Description: Four mutually exclusive categorical outcomes were defined based on the last valid Hamilton Depression Rating Scale (HDRS) rating at the Week 10 and Week 12 visits:
  1. Non-response: <30% reduction from baseline
  2. Partial Response: 30-49% reduction from baseline
  3. Response without remission: ≥50% reduction from baseline, but HDRS-17 score >7
  4. Remission: HDRS score ≤7
Time Frame: Measured at Weeks 10 and 12
Population: This population includes participants who completed the trial, per study protocol.
Measure: Number; unit: participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 86 | 79 | 69
participants
  Non-Response | 15 | 10 | 15
  Partial Response | 10 | 12 | 13
  Response without remission | 23 | 16 | 11
  Remission | 38 | 41 | 30

5. Secondary Outcome: Number of Participants Experiencing Depression Recurrence Following Remission to Monotherapy Treatment
Description: The number of participants experiencing a recurrence of depression after they had been in remission with the monotherapy treatment they were randomized to receive.
Time Frame: Measured at 6, 9, 12, 15, 18, 21, and 24 months
Population: This population is comprised of participants who completed 12 weeks of treatment, achieved remission, and participated in a follow-up phase that lasted for up to 21 months or until recurrence occurred.
Measure: Number; unit: participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 34 | 38 | 24
participants
  6 Months | 0 | 0 | 1
  9 Months | 1 | 2 | 1
  12 Months | 1 | 2 | 3
  15 Months | 1 | 4 | 5
  18 Months | 2 | 4 | 5
  21 Months | 3 | 5 | 5
  24 Months | 3 | 5 | 5

6. Secondary Outcome: Number of Participants Achieving Remission From Major Depressive Episode After 12 Weeks of Combined Treatment, for Those Patients Who do Not Achieve Remission With Monotherapy
Description: The number of participants achieving remission from major depressive episode after 12 weeks of combined treatment consisting of antidepressant plus cognitive behavioral therapy (CBT) treatments. Those originally randomized to receive one of the antidepressants remained on that medication and had CBT sessions added. Participants originally randomized to CBT had escitalopram added at a dose of 10 to 20 mg per day for 12 weeks
Time Frame: Measured after 12 weeks of combined treatment
Population: Participants who did not achieve remission during monotherapy were offered 12 weeks of combination therapy. This sample consists of those participants who consented for the combination therapy part of the trial and who completed the 12 weeks of treatment.
Measure: Number; unit: participants
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 41 | 25 | 31
participants | 22 | 10 | 18

ADVERSE EVENTS:
Time Frame: Adverse events will be collected during the entire time a participant remains in the trial (up to 24 weeks)
Arm/Group | Escitalopram | Duloxetine | Cognitive Behavioral Therapy (CBT)
Serious Adverse Events (participants affected / at risk) | 6/114 | 3/115 | 1/115
Other Adverse Events (participants affected / at risk) | 100/114 | 108/115 | 70/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=114) | Duloxetine (N=115) | Cognitive Behavioral Therapy (CBT) (N=115)
Hospitalization for asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Motor Vehicle Accident (General disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
AttemptedSuicide by Overdose (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=114) | Duloxetine (N=115) | Cognitive Behavioral Therapy (CBT) (N=115)
Headache (General disorders) | 36 | 38 | 19
Nausea (Gastrointestinal disorders) | 29 | 37 | 8
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 14 | 31 | 27
Diarrhea (Gastrointestinal disorders) | 23 | 22 | 11
Fatigue (General disorders) | 22 | 27 | 2
Insomnia (General disorders) | 20 | 26 | 3
Dry Mouth (General disorders) | 18 | 28 | 2
Dizziness (General disorders) | 16 | 21 | 4
Sedation (General disorders) | 15 | 18 | 4
Abdominal Pain (Gastrointestinal disorders) | 7 | 13 | 7
Dyspepsia (Gastrointestinal disorders) | 9 | 10 | 6
Decreased Libido (Reproductive system and breast disorders) | 12 | 11 | 2
Constipation (Gastrointestinal disorders) | 9 | 13 | 2
Anxiety (Psychiatric disorders) | 9 | 10 | 3
Anorgasmia (Reproductive system and breast disorders) | 12 | 7 | 2
Yawning (General disorders) | 7 | 10 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 9 | 1
Bruxism (General disorders) | 8 | 6 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 3
Flatulence (Gastrointestinal disorders) | 6 | 5 | 3
Somnolence (General disorders) | 8 | 5 | 1
Feeling Jittery (General disorders) | 6 | 7 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 9 | 0
Abnormal Orgasm (Reproductive system and breast disorders) | 3 | 9 | 1
Blurred Vision (Eye disorders) | 6 | 4 | 2
Emotional Poverty (Psychiatric disorders) | 9 | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 7 | 1 | 1
Palpitations (Cardiac disorders) | 2 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes